CLINICAL TRIAL: NCT01554618
Title: A Phase 3, Double-Blind, Placebo-Controlled, Randomized, Multi-Center Study to Assess the Safety and Efficacy of Exenatide Once Weekly in Adolescents With Type 2 Diabetes
Brief Title: Safety and Efficacy Study of Exenatide Once Weekly in Adolescents With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5551C00002
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-10

CONDITIONS: Children and Adolescent With Type 2 Diabetes
Keywords: exenatide; type 2 diabetes; GLP-1 receptor agonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EQW (Experimental): Exenatide once weekly
  Interventions: Drug: Exenatide Once Weekly
- Placebo (Placebo Comparator): Placebo once weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide Once Weekly — 2 mg exenatide once weekly
  Other Names: BYDUREON
  Arms: EQW
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study examines the Safety and efficacy study of exenatide once weekly in children and adolescents with type 2 diabetes

DETAILED DESCRIPTION:
This Phase 3, double-blind (controlled assessment period), randomized, multicenter, placebo-controlled parallel study is designed to examine the efficacy and safety of EQW compared to placebo (PBO) in adolescents with type 2 diabetes for 24 weeks. This study will assess safety and efficacy of EQW (as monotherapy and adjunctive therapy to oral antidiabetic agents and/or insulin). At least 40% and not more than 60% of the randomized patients must be females. At least 40% of patients should be recruited from areas with similar ethnicity and lifestyle to those of the European Union member states. Long term safety and efficacy of EQW will subsequently be monitored for 28 weeks in the open-label, uncontrolled extension period (through Week 52). The study will be terminated at Visit 11 (Week 62/Study Termination) which will be a follow-up visit occurring 10 weeks after the last dose administration at Visit 10 (Week 52). This study will be conducted in 77 patients with type 2 diabetes treated with diet and exercise alone or in combination with a stable dose of oral antidiabetic agents and/or insulin for at least 2 months prior to screening. During the controlled assessment period, approximately 77 patients will be randomly assigned in a 5:2 ratio to either EQW 2 mg (Group A) or PBO (Group B), to yield at least 70 evaluable patients: at least 50 patients in the exenatide and at least 20 patients in the PBO group. Following the 24-week controlled assessment period, patients assigned to the EQW 2 mg treatment (Group A) will continue to be treated with EQW 2 mg during the extension period (through Week 52). Patients randomized to PBO (Group B) will receive EQW 2 mg beginning at the start of the extension period, Week 25 through Week 52. In addition to receiving study medications, all patients will participate in a lifestyle intervention program encompassing diet and physical activity modifications following the signing of the informed consent and assent forms (Visit 1 [Week -2]) through the end of the extension period (Week 52). Following Visit 11 (Week 62/Study Termination), patients whose height increase is at least 5 mm between Visit 8 (Week 28) and Visit 11 (Week 62/Study Termination) will participate in a long-term safety follow-up period. Patients who discontinue study medication prior to Visit 11 (Week 62/Study Termination) will also participate in the Extended Safety Follow-up Period, unless they have a height increase of less than 5 mm over a 6-month interval at study site visits prior to discontinuation of study medication. Patients who do not have height assessments at study-site visits over a 6-month interval prior to discontinuation of study medication will enter the Extended Safety Follow-up Period. The Extended Safety Follow Up Period will continue for up to 3 years or until the difference between two 6-month interval visits is less than a 5 mm increase (whichever comes first). No study medication will be administered during the Extended Safety Follow-up Period. Blood samples will be collected for calcitonin and carcinoembryonic antigen (CEA) laboratory measurements.

ELIGIBILITY:
Each patient must meet the following criteria to be enrolled in this study.

1. Is a child or an adolescent of 10 to <18 years old, at Visit 1 (Screening)
2. Has been diagnosed with type 2 diabetes mellitus per American Diabetes Association diagnostic criteria
3. HbA1c of 6.5% to 11.0%, inclusive, in patients not taking insulin/SU, and of 6.5% to 12.0%, inclusive, in patients taking insulin/SU, at Visit 1 (Screening)
4. Has a C-peptide of >0.6 ng/L at Visit 1 (Screening)
5. Has been treated with diet and exercise alone or in combination with a stable dose of an oral antidiabetic agent (e.g., metformin and/or SU) and/or insulin for their type 2 diabetes for at least 2 months prior to Visit 1 (Screening)
6. Has a fasting plasma glucose concentration <280 mg/dL (15.5 mmol/L) at Visit 1 (Screening)

Patients who meet any of the following criteria will be excluded from the study.

1. Has a clinically significant medical condition that could potentially affect study participation and/or personal well-being, as judged by the Investigator, including but not limited to the following conditions:

   1. Hepatic disease (defined by aspartate or alanine transaminase >3.0 times the upper limit of normal (ULN)
   2. Renal disease or serum creatinine >1.5 mg/dL (132.6 µmol/L) (males) or 1.4 mg/dL (123.8 µmol/L) (females)
   3. Gastrointestinal disease deemed significant by the Investigator
   4. Organ transplantation
   5. Chronic infection (e.g., tuberculosis, human immunodeficiency virus, hepatitis B virus, or hepatitis C virus)
   6. Clinically significant malignant disease (with the exception of basal and squamous cell carcinoma of the skin) within 5 years of Visit 1 (Screening)
2. Has positive antibody titers to glutamic acid decarboxylase (GAD65) or islet cell antigen (ICA512) at Visit 1 (Screening)
3. Has a personal or family history of elevated calcitonin, calcitonin >100 ng/L, medullary thyroid carcinoma, or multiple endocrine neoplasia-2
4. Has ever used exenatide (exenatide once weekly [exenatide LAR], exenatide BID, BYETTA, or any other formulation) or any glucagon-like peptide-1 (GLP-1) receptor agonist (e.g., liraglutide [Victoza®])
5. Is pregnant

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2011-12-02 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2021-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (16):
  - Research Site, Los Angeles, California
  - Research Site, New Haven, Connecticut
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Jackson, Mississippi
  - Research Site, Buffalo, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Rapid City, South Dakota
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Bulgaria (2):
  - Research Site, Pleven
  - Research Site, Sevlievo
- Hungary (3):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Szeged
- Israel (3):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Ramat Gan
- Research Site, Kuwait City, Kuwait
- Mexico (4):
  - Research Site, Aguascalientes
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Veracruz
- Ukraine (4):
  - Research Site, Chernivts?
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Odesa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Tamborlane WV, Bishai R, Geller D, Shehadeh N, Al-Abdulrazzaq D, Vazquez EM, Karoly E, Troja T, Doehring O, Carter D, Monyak J, Sjostrom CD. Once-Weekly Exenatide in Youth With Type 2 Diabetes. Diabetes Care. 2022 Aug 1;45(8):1833-1840. doi: 10.2337/dc21-2275. PMID 35679098
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5551C00002&attachmentIdentifier=0bc86ca3-7a75-4e8f-a9ad-4e5eecc559f2&fileName=D5551C00002_SAP_redacted.pdf&versionIdentifier=
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5551C00002&attachmentIdentifier=db17e8c6-3fcb-4682-a3b7-55f643581f58&fileName=D5551C00002_CSP_redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5551C00002&attachmentIdentifier=32faa63c-a8de-4c1a-9aa4-6a3c46170eef&fileName=D5551C00002_CSR_synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in adolescents (aged 10 to 17 years inclusive) with type 2 diabetes treated with diet and exercise alone or in combination with a stable dose of oral antidiabetic agents and/or insulin for at least 2 months prior to screening. 27 study centers in 6 countries randomized patients during the study.
Pre-assignment Details: Study had a screening period (5 weeks), controlled assessment period (24 weeks; patients randomized 5:2 to exenatide or placebo), open-label extension period (28 weeks) and post-treatment follow-up period (10 weeks). 84 patients were randomized but 1 due to clinical error and immediately discontinued, thus, 83 patients were included in the study.
Groups:
- Exenatide: Controlled assessment Period: Patients received exenatide 2 milligrams (mg) subcutaneous (SC) injection once weekly for 24 weeks.
  Extension period: Patients continued to receive exenatide 2 mg SC once weekly during the open-label extension period for 28 weeks (through Week 52).
- Placebo: Controlled assessment period: Patients received placebo (matching with exenatide) SC injection once weekly for 24 weeks.
  Extension period: Patients then received exenatide 2 mg SC once weekly beginning at the start of the open-label extension period for 28 weeks (from Week 25 to Week 52).
Period: Randomized Through Start of Treatment
Arm/Group | Exenatide | Placebo
Started | 59 | 24
Completed | 58 | 24
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Controlled Assessment Period
Arm/Group | Exenatide | Placebo
Started (Received treatment during controlled assessment period) | 58 | 24
Completed (Completed controlled assessment period) | 50 | 23
Not Completed | 8 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 6 | 0
Period: Open-Label Extension Period
Arm/Group | Exenatide | Placebo
Started (Received open-label exenatide treatment) | 49 (1 patient who was noncompliant with study medication did not enter the open-label extension period) | 23
Completed (Completed extension period) | 46 | 18
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis performed on Intent-to-Treat (ITT) Analysis Set which consisted of all randomized patients who received at least 1 dose of randomized study medication.
Groups:
- Exenatide: Controlled assessment period: Patients received exenatide 2 mg SC injection once weekly for 24 weeks.
  Extension period: Patients continued to receive exenatide 2 mg SC once weekly during the open-label extension period for 28 weeks (through Week 52).
- Total: Total of all reporting groups
Arm/Group | Exenatide | Placebo | Total
Number analyzed (Participants) | 58 | 24 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (1.88) | 15.6 (1.66) | 15.1 (1.84)
Age, Customized [Count of Participants; unit: Participants] — Age group (years)
  Participants
    < 10 | 0 | 0 | 0
    ≥ 10 to ≤ 12 | 8 | 3 | 11
    ≥ 13 to ≤ 16 | 36 | 12 | 48
    > 16 | 14 | 9 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 17 | 48
  Male | 27 | 7 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 8 | 33
  Not Hispanic or Latino | 29 | 13 | 42
  Unknown or Not Reported | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 12 | 35
  Black or African American | 17 | 8 | 25
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 4 | 1 | 5
  Other | 12 | 2 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 1 | 0 | 1
  Hungary | 3 | 1 | 4
  Israel | 4 | 3 | 7
  Mexico | 13 | 2 | 15
  United States | 35 | 17 | 52
  Kuwait | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) to Week 24 (Controlled Assessment Period)
Description: Change from baseline in HbA1c (%) to Week 24 during the controlled assessment period is reported as adjusted least square (LS) mean values. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. A mixed model with repeated measures (MMRM) analysis was performed, excluding data collected after initiation of rescue medication or premature discontinuation of study medication.
Time Frame: Baseline (Week 0) and Week 24
Population: The Evaluable Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication and had at least 1 baseline and post-baseline HbA1c assessment.
Measure: Least Squares Mean (Standard Error); unit: percentage (% HbA1c)
Groups:
- Controlled Assessment Period - Exenatide: Patients received exenatide 2 mg SC injection once weekly for 24 weeks during the controlled assessment period.
- Controlled Assessment Period - Placebo: Patients received placebo (matching with exenatide) SC injection once weekly for 24 weeks during the controlled assessment period.
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 58 | 24
percentage (% HbA1c) | -0.36 (0.184) | 0.49 (0.273)
Statistical Analysis 1: Comparison: Controlled Assessment Period - Placebo; Adjusted LS mean and treatment group difference in the change from baseline at Week 24 were modeled using a MMRM including treatment group, region, visit, and treatment group by visit interaction, baseline HbA1c value (continuous) and baseline HbA1c by visit interaction as fixed effects, using an unstructured covariance matrix; Test type: Superiority; p = 0.012, Mixed Models Analysis; LS Mean Difference = -0.85, 95% CI 2-sided [-1.51 to -0.19], Standard Error of Mean 0.330 — Exenatide versus Placebo

2. Primary Outcome: Percentage of Patients With On-Treatment Adverse Events (AEs) up to Week 24 (Controlled Assessment Period)
Description: A controlled assessment period AE was defined as an AE starting on or after day of first dose of study medication up to but not including Week 24 for patients entering the extension period. For patients not entering the extension period, the period was defined up to and including last dose of study medication + 7 days (+ 90 days for serious AEs [SAEs] and other clinically significant or related AEs). The Investigator assessed AEs for causal relationship to study drug medication.
Time Frame: Day 1 (Week 0) up to Week 24, plus up to a maximum of 90 days follow up
Population: The Safety Analysis Set consisted of all patients who received at least 1 dose of study medication. One patient who was randomized to placebo received a dose of exenatide in error and was subsequently reassigned to the exenatide treatment group for analyses based on actual treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 59 | 23
percentage of participants
  Any AE | 61.0 | 73.9
  Any AE with outcome of death | 0 | 0
  Any SAE | 3.4 | 4.3
  Any AE leading to discontinuation of treatment | 0 | 0
  Any AE leading to discontinuation from study | 0 | 0
  Any AE related to treatment | 25.4 | 21.7

3. Primary Outcome: Percentage of Patients Positive for Anti-Drug Antibodies (ADAs) to Exenatide up to Week 24
Description: Percentage of patients positive for ADAs up to Week 24 for the exenatide treatment group is reported. Baseline was the antibody measurement at Week 0 (Day 1). A negative or missing antibody measurement was considered negative at baseline. High positive = antibody titers ≥ 625, including baseline assessment. Low positive = antibody titers < 625, including baseline assessment. A patient was said to have treatment-emergent ADA positive at a visit if the antibody test was positive after the first dose of exenatide following a negative or missing antibody measurement, or the titer increased by at least 1 titration category from a detectable measurement prior to first dose of randomized study medication.
Time Frame: Samples were collected on Day 1 (Week 0), Week 4, Week 8, Week 12 and Week 24
Population: The Safety Analysis Set consisted of all patients who received at least 1 dose of study medication. Only patients receiving exenatide in the controlled assessment period were included in the analysis.
Measure: Number; unit: percentage of participants
Groups:
- Treatment Period - Exenatide: Patients received exenatide 2 mg SC injection once weekly for 24 weeks during the controlled assessment period and continued to receive exenatide 2 mg SC once weekly during the open-label extension period for a further 28 weeks (from Week 0 to Week 52 overall).
Arm/Group | Treatment Period - Exenatide
Number analyzed (Participants) | 59
percentage of participants
  Week 4: High Positive: number analyzed (Participants) | 53
  Week 4: High Positive | 17.0
  Week 4: Low Positive: number analyzed (Participants) | 53
  Week 4: Low Positive | 30.2
  Week 4: Treatment-Emergent ADA Positive: number analyzed (Participants) | 53
  Week 4: Treatment-Emergent ADA Positive | 45.3
  Week 8: High Positive: number analyzed (Participants) | 52
  Week 8: High Positive | 53.8
  Week 8: Low Positive: number analyzed (Participants) | 52
  Week 8: Low Positive | 38.5
  Week 8: Treatment-Emergent ADA Positive: number analyzed (Participants) | 52
  Week 8: Treatment-Emergent ADA Positive | 92.3
  Week 12: High Positive: number analyzed (Participants) | 50
  Week 12: High Positive | 60.0
  Week 12: Low Positive: number analyzed (Participants) | 50
  Week 12: Low Positive | 38.0
  Week 12: Treatment-Emergent ADA Positive: number analyzed (Participants) | 50
  Week 12: Treatment-Emergent ADA Positive | 98.0
  Week 24: High Positive: number analyzed (Participants) | 49
  Week 24: High Positive | 40.8
  Week 24: Low Positive: number analyzed (Participants) | 49
  Week 24: Low Positive | 55.1
  Week 24: Treatment-Emergent ADA Positive: number analyzed (Participants) | 49
  Week 24: Treatment-Emergent ADA Positive | 95.9

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) Concentration to Week 24 (Controlled Assessment Period)
Description: Change from baseline in FPG to Week 24 during the controlled assessment period is reported as adjusted LS mean values. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. A MMRM analysis was performed, excluding data collected after initiation of rescue medication or after premature discontinuation of study medication.
Time Frame: Baseline (Week 0) and Week 24
Population: The ITT Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 58 | 24
milligrams per deciliter (mg/dL) | -5.2 (7.65) | 16.5 (11.32)
Statistical Analysis 1: Comparison: Controlled Assessment Period - Placebo; Adjusted LS mean and treatment group difference in the change from baseline at Week 24 were modeled using a MMRM including treatment group, region, visit, and treatment group by visit interaction, baseline fasting plasma glucose value, screening HbA1c (< 9.0% or ≥ 9.0%), and baseline fasting plasma glucose by visit interaction as fixed effects, using an unstructured covariance matrix; Test type: Superiority; p = 0.119, Mixed Models Analysis; LS Mean Difference = -21.6, 95% CI 2-sided [-49.0 to 5.7], Standard Error of Mean 13.70 — Exenatide versus Placebo

5. Secondary Outcome: Change From Baseline in Body Weight to Week 24 (Controlled Assessment Period)
Description: Change from baseline in body weight to Week 24 during the controlled assessment period is reported as adjusted LS mean values. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. A MMRM analysis was performed, excluding data collected after initiation of rescue medication or after premature discontinuation of study medication.
Time Frame: Baseline (Week 0) and Week 24
Population: The ITT Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 58 | 24
kilogram (kg) | -0.59 (0.665) | 0.63 (0.982)
Statistical Analysis 1: Comparison: Controlled Assessment Period - Placebo; Adjusted LS mean and treatment group difference in the change from baseline at Week 24 were modeled using a MMRM including treatment group, region, visit, and treatment group by visit interaction, baseline body weight, screening HbA1c (< 9.0% or ≥ 9.0%), and baseline body weight by visit interaction as fixed effects, using an unstructured covariance matrix; Test type: Superiority; p = 0.307, Mixed Models Analysis; LS Mean Difference = -1.22, 95% CI 2-sided [-3.59 to 1.15], Standard Error of Mean 1.189 — Exenatide versus Placebo

6. Secondary Outcome: Change From Baseline in Fasting Insulin to Week 24 (Controlled Assessment Period)
Description: Change from baseline in fasting insulin to Week 24 during the controlled assessment period is reported as adjusted LS mean values. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. A MMRM analysis was performed, excluding data collected after initiation of rescue medication or after premature discontinuation of study medication.
Time Frame: Baseline (Week 0) and Week 24
Population: The ITT Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication.
Measure: Least Squares Mean (Standard Error); unit: picomoles per liter (pmol/L)
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 58 | 24
picomoles per liter (pmol/L) | 79.6 (52.28) | -15.3 (78.49)
Statistical Analysis 1: Comparison: Controlled Assessment Period - Placebo; Adjusted LS mean and treatment group difference in the change from baseline at Week 24 were modeled using a MMRM including treatment group, region, visit, treatment group by visit interaction, baseline fasting insulin, screening HbA1c (< 9.0% or ≥ 9.0%), and baseline fasting insulin by visit interaction as fixed effects, using an unstructured covariance matrix; Test type: Superiority; p = 0.323, Mixed Models Analysis; LS Mean Difference = 94.9, 95% CI 2-sided [-95.6 to 285.5], Standard Error of Mean 95.26 — Exenatide versus Placebo

7. Secondary Outcome: Percentage of Patients Achieving HbA1c Goals of < 6.5%, ≤ 6.5%, and < 7.0% at Week 24 (Controlled Assessment Period)
Description: The percentage of patients achieving HbA1c goals of < 6.5%, ≤ 6.5%, and < 7.0% at Week 24 during the controlled assessment period is reported. A Cochran-Mantel-Haenszel (CMH) analysis was performed with missing data treated as non-responder, and excluding data collected after initiation of rescue medication or after premature discontinuation of study medication.
Time Frame: At Week 24
Population: The Evaluable Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication and had at least 1 baseline and post-baseline HbA1c assessment. Only patients with data available were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 48 | 22
percentage of participants
  HbA1c <6 .5% | 19.0 [8.9 to 29.1] | 4.2 [0.0 to 12.2]
  HbA1c ≤ 6.5% | 19.0 [8.9 to 29.1] | 4.2 [0.0 to 12.2]
  HbA1c < 7.0% | 31.0 [19.1 to 42.9] | 8.3 [0.0 to 19.4]
Statistical Analysis 1: Comparison: Controlled Assessment Period - Placebo; Treatment difference in HbA1c < 6.5%: Treatment group comparison was based on CMH test stratified by screening HbA1c (<9.0% or >=9.0%). P-value was from the general association statistic; Test type: Superiority; p = 0.077, Cochran-Mantel-Haenszel; Difference = 14.8, 95% CI 2-sided [1.9 to 27.7] — Exenatide versus Placebo. Difference was the risk difference of the 2 proportions
Statistical Analysis 2: Comparison: Controlled Assessment Period - Placebo; Treatment difference in HbA1c ≤ 6.5%: Treatment group comparison was based on CMH test stratified by screening HbA1c (<9.0% or >=9.0%). P-value was from the general association statistic; Test type: Superiority; p = 0.077, Cochran-Mantel-Haenszel; Difference = 14.8, 95% CI 2-sided [1.9 to 27.7] — Exenatide versus Placebo. Difference was the risk difference of the 2 proportions
Statistical Analysis 3: Comparison: Controlled Assessment Period - Placebo; Treatment difference in HbA1c < 7.0%: Treatment group comparison was based on CMH test stratified by screening HbA1c (<9.0% or >=9.0%). P-value was from the general association statistic; Test type: Superiority; p = 0.020, Cochran-Mantel-Haenszel; Difference = 22.7, 95% CI 2-sided [6.5 to 39.0] — Exenatide versus Placebo. Difference was the risk difference of the 2 proportions

8. Secondary Outcome: Change From Baseline in Lipid Profiles to Week 24 (Controlled Assessment Period)
Description: Change from baseline in lipid profiles to Week 24 during the controlled assessment period is reported as mean values (Standard International [SI] units). The following lipids were assessed: total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and triglycerides. All lipids presented were taken in a fasted state. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. Data collected after initiation of rescue medication or after premature discontinuation of study medication were excluded.
Time Frame: Baseline (Week 0) and Week 24
Population: The ITT Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication. Only patients with data available were included in the analysis.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 58 | 24
millimoles per liter (mmol/L)
  Total Cholesterol: number analyzed (Participants) | 46 | 21
  Total Cholesterol | -0.117 (0.7124) | -0.114 (0.5819)
  HDL-C: number analyzed (Participants) | 46 | 21
  HDL-C | -0.035 (0.1950) | -0.047 (0.1039)
  LDL-C: number analyzed (Participants) | 43 | 20
  LDL-C | -0.050 (0.5618) | -0.110 (0.5983)
  Triglycerides: number analyzed (Participants) | 46 | 21
  Triglycerides | -0.122 (1.0303) | 0.094 (0.6626)

9. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) to Week 24 (Controlled Assessment Period)
Description: Change from baseline in SBP and DBP to Week 24 during the controlled assessment period is reported as adjusted LS mean values. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. A MMRM analysis was performed, excluding data collected after initiation of rescue medication or after premature discontinuation of study medication.
Time Frame: Baseline (Week 0) and Week 24
Population: The ITT Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication.
Measure: Least Squares Mean (Standard Error); unit: millimeters mercury (mmHg)
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 58 | 24
millimeters mercury (mmHg)
  SBP | -0.7 (1.48) | 2.2 (2.15)
  DBP | 0.2 (1.00) | -1.3 (1.45)
Statistical Analysis 1: Comparison: Controlled Assessment Period - Placebo; Treatment difference in SBP: Adjusted LS mean and treatment group difference in the change from baseline at Week 24 were modeled using a MMRM including treatment group, region, visit, treatment group by visit interaction, baseline SBP, screening HbA1c (< 9.0% or ≥ 9.0%), and baseline SBP by visit interaction as fixed effects, using an unstructured covariance matrix; Test type: Superiority; p = 0.284, Mixed Models Analysis; LS Mean Difference = -2.8, 95% CI 2-sided [-8.0 to 2.4], Standard Error of Mean 2.61 — Exenatide versus Placebo
Statistical Analysis 2: Comparison: Controlled Assessment Period - Placebo; Treatment difference in DBP: Adjusted LS mean and treatment group difference in the change from baseline at Week 24 were modeled using a MMRM including treatment group, region, visit, treatment group by visit interaction, baseline DBP, screening HbA1c (< 9.0% or ≥ 9.0%), and baseline DBP by visit interaction as fixed effects, using an unstructured covariance matrix; Test type: Superiority; p = 0.376, Mixed Models Analysis; LS Mean Difference = 1.6, 95% CI 2-sided [-2.0 to 5.1], Standard Error of Mean 1.77 — Exenatide versus Placebo

10. Secondary Outcome: Number of Patients Needing Rescue Medication Due to Failure to Maintain Glycemic Control up to Week 24 (Controlled Assessment Period)
Description: Number of patients needing rescue medication at Week 24 and at each intermediate visit during the controlled assessment period is reported. Patients with a loss of glycemic control, defined as either an increase from baseline in HbA1c values by ≥ 1.0% at 2 consecutive clinic visits that were at least 1 month apart, or a fasting plasma glucose value ≥ 250 mg/dL or random blood glucose value > 300 mg/dL for 4 days during a 7 day period, received rescue medication. Data collected after premature discontinuation of study medication were excluded.
Time Frame: At Week 4, Week 8, Week 12, Week 18 and Week 24
Population: The ITT Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication. Only patients with data available at each specified visit were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 58 | 24
Participants
  Week 4: number analyzed (Participants) | 57 | 24
  Week 4 | 0 | 0
  Week 8: number analyzed (Participants) | 55 | 24
  Week 8 | 0 | 0
  Week 12: number analyzed (Participants) | 51 | 24
  Week 12 | 0 | 0
  Week 18: number analyzed (Participants) | 50 | 24
  Week 18 | 1 | 0
  Week 24: number analyzed (Participants) | 49 | 24
  Week 24 | 0 | 0

11. Secondary Outcome: Change From Baseline in Homeostasis Model Assessments - Beta-Cell Function (HOMA-B) and Insulin Sensitivity (HOMA-S) to Week 24 (Controlled Assessment Period)
Description: Change from baseline in HOMA-B and HOMA-S in patients who were not taking insulin to Week 24 during the controlled assessment period is reported as adjusted LS mean values. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. A MMRM analysis was performed, excluding data collected after initiation of rescue medication or after premature discontinuation of study medication.
Time Frame: Baseline (Week 0) and Week 24
Population: The ITT Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication. Homeostasis model assessments were only performed in patients who were not taking insulin.
Measure: Least Squares Mean (Standard Error); unit: percentage (%HOMA-B and %HOMA-S)
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 14 | 7
percentage (%HOMA-B and %HOMA-S)
  HOMA-B | 63.98 (39.552) | -26.39 (56.138)
  HOMA-S | 0.62 (3.607) | 7.37 (4.914)
Statistical Analysis 1: Comparison: Controlled Assessment Period - Placebo; Treatment difference in HOMA-B: Adjusted LS mean and treatment group difference in the change from baseline at Week 24 were modeled using a MMRM including treatment group, region, visit, treatment group by visit interaction, baseline HOMA-B, screening HbA1c (< 9.0% or ≥ 9.0%), and baseline HOMA-B by visit interaction as fixed effects, using an unstructured covariance matrix; Test type: Superiority; p = 0.211, Mixed Models Analysis; LS Mean Difference = 90.37, 95% CI 2-sided [-57.27 to 238.00], Standard Error of Mean 69.207 — Exenatide versus Placebo
Statistical Analysis 2: Comparison: Controlled Assessment Period - Placebo; Treatment difference in HOMA-S: Adjusted LS mean and treatment group difference in the change from baseline at Week 24 were modeled using a MMRM including treatment group, region, visit, treatment group by visit interaction, baseline HOMA-S, screening HbA1c (< 9.0% or ≥ 9.0%), and baseline HOMA-S by visit interaction as fixed effects, using an unstructured covariance matrix; Test type: Superiority; p = 0.289, Mixed Models Analysis; LS Mean Difference = -6.75, 95% CI 2-sided [-19.80 to 6.29], Standard Error of Mean 6.173 — Exenatide versus Placebo

12. Secondary Outcome: Percentage of Patients Reporting AEs of Injection Site Reactions up to Week 24 (Controlled Assessment Period)
Description: Percentage of patients reporting injection site reactions at Week 24 and at each intermediate visit during the controlled assessment period is reported. Injection site reactions were presented from the AE case report form (CRF), based on the "Injection site reactions" higher level term. A controlled assessment period AE was defined as an AE starting on or after day of first dose of study medication up to but not including Week 24 for patients entering the extension period. For patients not entering the extension period, the period was defined up to and including last dose of study medication + 7 days (+ 90 days for SAEs and other clinically significant or related AEs).
Time Frame: At Week 4, Week 8, Week 12, Week 18 and Week 24
Population: The Safety Analysis Set consisted of all patients who received at least 1 dose of study medication. Only patients with data available at each specified visit were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo
Number analyzed (Participants) | 59 | 23
percentage of participants
  Week 4 | 8.5 | 8.7
  Week 8: number analyzed (Participants) | 57 | 23
  Week 8 | 3.5 | 4.3
  Week 12: number analyzed (Participants) | 53 | 23
  Week 12 | 1.9 | 0
  Week 18: number analyzed (Participants) | 51 | 22
  Week 18 | 0 | 0
  Week 24: number analyzed (Participants) | 51 | 22
  Week 24 | 0 | 0

13. Secondary Outcome: Change From Baseline in HbA1c to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: Change from baseline in HbA1c (%) to Week 52 among patients who received open-label exenatide during the treatment period is reported as mean values. The treatment period was defined as the controlled assessment period and extension period combined. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. Data collected after initiation of rescue medication or after premature discontinuation of study medication were excluded.
Time Frame: Baseline (Week 0) and Week 52
Population: The Evaluable Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication and had at least 1 baseline and post-baseline HbA1c assessment. Only patients with observed baseline and Week 52 values, and who received open-label exenatide were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage (% HbA1c)
Groups:
- Treatment Period - Placebo Then Exenatide: Patients received placebo (matching with exenatide) SC injection once weekly for 24 weeks during the controlled assessment period and then received exenatide 2 mg SC once weekly beginning at the start of the open-label extension period for 28 weeks (from Week 25 to Week 52).
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 39 | 17
percentage (% HbA1c) | -0.10 (1.711) | 0.53 (2.123)

14. Secondary Outcome: Change From Baseline in FPG Concentration to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: Change from baseline in FPG to Week 52 among patients who received open-label exenatide during the treatment period is reported as mean values. The treatment period was defined as the controlled assessment period and extension period combined. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. Data collected after initiation of rescue medication or after premature discontinuation of study medication were excluded.
Time Frame: Baseline (Week 0) and Week 52
Population: The ITT Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication. Only patients with observed baseline and Week 52 values, and who received open-label exenatide were included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 38 | 16
mg/dL | -1.8 (62.64) | 10.6 (75.49)

15. Secondary Outcome: Change From Baseline in Body Weight to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: Change from baseline in body weight to Week 52 among patients who received open-label exenatide during the treatment period is reported as mean values. The treatment period was defined as the controlled assessment period and extension period combined. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. Data collected after initiation of rescue medication or after premature discontinuation of study medication were excluded.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 39 | 18
kg | 0.04 (6.088) | -0.04 (4.687)

16. Secondary Outcome: Change From Baseline in Fasting Insulin to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: Change from baseline in fasting insulin to Week 52 among patients who received open-label exenatide during the treatment period is reported as mean values. The treatment period was defined as the controlled assessment period and extension period combined. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. Data collected after initiation of rescue medication or after premature discontinuation of study medication were excluded.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 37 | 16
pmol/L | -32.4 (273.57) | 121.5 (379.13)

17. Secondary Outcome: Percentage of Participants Achieving HbA1c Goals of < 6.5%, ≤ 6.5%, and < 7.0% to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: The percentage of patients achieving HbA1c goals of < 6.5%, ≤ 6.5%, and < 7.0% at Week 52 among patients who received open-label exenatide during the treatment period is reported. The treatment period was defined as the controlled assessment period and extension period combined. Data collected after initiation of rescue medication or after premature discontinuation of study medication were excluded.
Time Frame: At Week 52
Population: The Evaluable Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication and had at least 1 baseline and post-baseline HbA1c assessment. Only patients who received open-label exenatide and with data available were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 39 | 17
percentage of participants
  HbA1c < 6.5% | 30.8 | 23.5
  HbA1c ≤ 6.5% | 30.8 | 23.5
  HbA1c < 7.0% | 35.9 | 29.4

18. Secondary Outcome: Change From Baseline in Lipids Profiles to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: Change from baseline in lipid profiles to Week 52 among patients who received open-label exenatide during the treatment period is reported as mean values (SI units). The treatment period was defined as the controlled assessment period and extension period combined. The following lipids were assessed: total cholesterol, HDL-C, LDL-C, and triglycerides. All lipids presented were taken in a fasted state. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. Data collected after initiation of rescue medication or after premature discontinuation of study medication were excluded.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 37 | 15
mmol/L
  Total Cholesterol | -0.188 (0.4199) | -0.255 (0.9075)
  HDL-C | 0.004 (0.1740) | -0.076 (0.2327)
  LDL-C: number analyzed (Participants) | 33 | 15
  LDL-C | -0.175 (0.4025) | -0.152 (0.7682)
  Triglycerides | -0.155 (1.1108) | -0.043 (0.5971)

19. Secondary Outcome: Change From Baseline in Blood Pressure (Systolic and Diastolic) to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: Change from baseline in SBP and DBP to Week 52 among patients who received open-label exenatide during the treatment period is reported as mean values. The treatment period was defined as the controlled assessment period and extension period combined. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. Data collected after initiation of rescue medication or after premature discontinuation of study medication were excluded.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 39 | 18
mmHg
  SBP | -0.7 (13.09) | -0.6 (8.73)
  DBP | 1.1 (8.65) | -2.5 (10.65)

20. Secondary Outcome: Number of Patients Needing Rescue Medication Due to Failure to Maintain Glycemic Control up to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: Number of patients needing rescue medication at Week 52 and at each intermediate visit during the treatment period is reported. The treatment period was defined as the controlled assessment period and extension period combined. Patients with a loss of glycemic control, defined as either an increase from baseline in HbA1c values by ≥ 1.0% at 2 consecutive clinic visits that were at least 1 month apart, or a fasting plasma glucose value ≥ 250 mg/dL or random blood glucose value > 300 mg/dL for 4 days during a 7 day period, received rescue medication. Data collected after premature discontinuation of study medication were excluded.
Time Frame: At Week 4, Week 8, Week 12, Week 18, Week 24, Week 28, Week 40 and Week 52
Population: The ITT Analysis Set consisted of all randomized patients who received at least 1 dose of randomized study medication. Only patients who received open-label exenatide and with data available were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 49 | 23
Participants
  Week 4 | 0 | 0
  Week 8 | 0 | 0
  Week 12 | 0 | 0
  Week 18 | 1 | 0
  Week 24 | 0 | 0
  Week 28 | 2 | 1
  Week 40: number analyzed (Participants) | 47 | 20
  Week 40 | 2 | 0
  Week 52: number analyzed (Participants) | 45 | 18
  Week 52 | 0 | 0

21. Secondary Outcome: Change From Baseline in HOMA-B and HOMA-S to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: Change from baseline in HOMA-B and HOMA-S to Week 52 among patients who received open-label exenatide during the treatment period is reported as mean values. The treatment period was defined as the controlled assessment period and extension period combined. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of randomized study medication. Data collected after initiation of rescue medication or after premature discontinuation of study medication were excluded.
Time Frame: Baseline (Week 0) and Week 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percentage (%HOMA-B and %HOMA-S)
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 8 | 5
percentage (%HOMA-B and %HOMA-S)
  HOMA-B | -2.58 (130.435) | 42.02 (183.869)
  HOMA-S | 9.85 (12.366) | 2.36 (7.631)

22. Secondary Outcome: Percentage of Patients Reporting AEs of Injection Site Reactions up to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: Percentage of patients reporting injection site reactions at Week 52 and at each intermediate visit among patients who received open-label exenatide during the treatment period is reported. The treatment period was defined as the controlled assessment period and extension period combined. Injection site reactions were presented from the AE CRF, based on the "Injection site reactions" higher level term. An Extension Period AE was defined as an AE starting on or after day of first dose of open-label exenatide to last dose + 7 days (+ 90 days for SAEs and other clinically significant or related AEs).
Time Frame: At Week 4, Week 8, Week 12, Week 18, Week 24, Week 28, Week 40 and Week 52
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 50 | 22
percentage of participants
  Week 4 | 10.0 | 9.1
  Week 8 | 4.0 | 4.5
  Week 12 | 2.0 | 0
  Week 18 | 0 | 0
  Week 24 | 0 | 0
  Week 28 | 4.0 | 0
  Week 40: number analyzed (Participants) | 48 | 19
  Week 40 | 0 | 0
  Week 52: number analyzed (Participants) | 46 | 17
  Week 52 | 0 | 0

23. Secondary Outcome: Plasma Exenatide Concentrations to Week 52 Among Patients Who Received Open-Label Exenatide (Treatment Period)
Description: Geometric mean plasma exenatide concentrations up to Week 52 during the treatment period are reported (for the placebo then exenatide treatment group, only Weeks 24 and 52 were applicable). The treatment period was defined as the controlled assessment period and extension period combined. Data collected after initiation of rescue medication were included. Data collected after discontinuation of study medication were excluded.
Time Frame: Samples were collected on Day 1 (Week 0), Week 4, Week 8, Week 12, Week 24 and Week 52
Population: The Pharmacokinetic (PK) Analysis Set consisted of all patients who received at least 1 dose of exenatide, for whom any postdose data were available and who did not deviate from the protocol in ways that would significantly affect the PK analyses. Only patients who received open-label exenatide and with data available were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter
Arm/Group | Treatment Period - Exenatide | Treatment Period - Placebo Then Exenatide
Number analyzed (Participants) | 55 | 19
picograms per milliliter
  Baseline: number analyzed (Participants) | 54 | 0
  Baseline | NA (NA) — Not calculated as below the lower limit of quantification. |
  Week 4: number analyzed (Participants) | 54 | 0
  Week 4 | 41.51 (91.9) |
  Week 8: number analyzed (Participants) | 49 | 0
  Week 8 | 130.60 (83.8) |
  Week 12: number analyzed (Participants) | 44 | 0
  Week 12 | 163.58 (92.3) |
  Week 24: number analyzed (Participants) | 33 | 18
  Week 24 | 140.81 (84.0) | NA (NA) — Not calculated as below the lower limit of quantification.
  Week 52: number analyzed (Participants) | 28 | 17
  Week 52 | 88.88 (79.2) | 105.56 (154.9)

ADVERSE EVENTS:
Time Frame: After the first dose of study medication in period through the end of the treatment in period + 90 days for SAEs (or + 7 days for non-serious (i.e. Other) AEs. Overall time frame: up to maximum of approximately 37 weeks and 41 weeks for controlled assessment period and extension period, respectively.
Description: The Safety Analysis Set consisted of all patients who received at least 1 dose of study medication. One patient who was randomized to placebo received a dose of exenatide in error and was subsequently reassigned to the exenatide treatment group for analyses based on actual treatment (ie, for analyses based on the Safety Analysis Set).
Groups:
- Extension Period - Exenatide: Patients received open-label exenatide 2 mg SC injection once weekly for 28 weeks during the extension period. Patients in this treatment group had previously received exenatide during the controlled assessment period.
- Extension Period - Placebo to Exenatide: Patients received open-label exenatide 2 mg SC injection once weekly for 28 weeks during the extension period. Patients in this treatment group had previously received placebo during the controlled assessment period.
Arm/Group | Controlled Assessment Period - Exenatide | Controlled Assessment Period - Placebo | Extension Period - Exenatide | Extension Period - Placebo to Exenatide
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/23 | 0/50 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/59 | 1/23 | 3/50 | 1/22
Other Adverse Events (participants affected / at risk) | 25/59 | 10/23 | 10/50 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Controlled Assessment Period - Exenatide (N=59) | Controlled Assessment Period - Placebo (N=23) | Extension Period - Exenatide (N=50) | Extension Period - Placebo to Exenatide (N=22)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Controlled Assessment Period - Exenatide (N=59) | Controlled Assessment Period - Placebo (N=23) | Extension Period - Exenatide (N=50) | Extension Period - Placebo to Exenatide (N=22)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 3 (3) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Injection site erythema (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 2 (3) | 1 (1) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 2 (3) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 0 (0) | 2 (3)

LIMITATIONS AND CAVEATS:
For statistical analyses of change from baseline in HOMA-B and HOMA-S, due to the limited sample size (n=14 and n=7 in the extenatide and placebo groups, respectively) it is difficult to accurately interpret these data. The study design included an extended safety follow-up period which continued for up to 3 years or until the increase in height between two 6-month interval visits was <5 mm (whichever came first). No study medication was administered during the extended safety follow-up period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT01554618/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT01554618/SAP_003.pdf